CLINICAL TRIAL: NCT05476094
Title: A Randomized, Double-blind, Placebo-controlled, Single Center and Single Dose Phase Ⅰ Study to Evaluate Pharmacokinetic/Pharmacodynamic Characteristics and Safety/Tolerability of AYP-101 S.C. Injection in Healthy Subjects
Brief Title: Evaluate Pharmacokinetic/Pharmacodynamic and Safety/Tolerability of AYP-101 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AMIpharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AYP-101-101
Record Dates: First submitted 2022-07-15; First posted 2022-07-27 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Healthy Subjects; Submental Fat
Keywords: submental fat
MeSH Terms: interventions — polyene phosphatidylcholine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A Randomized, Double-blind, Placebo-controlled, Single Center and Single Dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: AYP-101 1 (Experimental): 0.2 mL injections, 1.0 cm apart, up to 10.0 ml, Single administration
  Interventions: Drug: Polyene Phosphatidylcholine
- Experimental: AYP-101 2 (Experimental): 0.2 mL injections, 1.0 cm apart, up to 10.0 ml, Single administration
  Interventions: Drug: Polyene Phosphatidylcholine
- Placebo (Placebo Comparator): 0.2 mL injections, 1.0 cm apart, up to 10.0 ml, Single administration
  Interventions: Drug: Polyene Phosphatidylcholine

INTERVENTIONS:
Drug: Polyene Phosphatidylcholine — AYP-101 1 - 25 mg of essential phospholipids in 1 mL AYP-101 2 - 50 mg of essential phospholipids in 1 mL Placebo - Essential phospholipids in 1 mL 00 mg
  Other Names: AYP-101 1; AYP-101 2; Placebo

SUMMARY:
To Evaluate Pharmacokinetic/Pharmacodynamic Characteristics and Safety/Tolerability of AYP-101 S.C. injection in Healthy Subjects

A Randomized, Double-blind, Placebo-controlled, Single Center and Single Dose

DETAILED DESCRIPTION:
This study is planed to Evaluate Pharmacokinetic/Pharmacodynamic Characteristics and Safety/Tolerability of AYP-101 S.C. injection in Healthy Subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female equal to or greater than 19 and equal to or less than 65 years old
2. submental fat under the chin capable of a single S.C. injection - 50 points at intervals of 1.0 cm grid pattern (90% or more, i.e. a minimum of 45 points, if not enough points)
3. BMI(Body Mass Index, kg/m^2) - 19.0 or more and less than 35.0
4. agree to contraception through medically permitted contraceptive methods during clinical trial (three months after final administration) among potentially pregnant men and women
5. agree not to donate or transfuse blood (including whole blood, plasma components, platelet components, and platelet plasma components) during clinical trial
6. agree not to receive adiposeform therapy (fat inhalation, surgery, etc.) or cosmetic surgery (botox, filler, laser, high frequency, etc.) at other sites of administration during clinical trial
7. Singed informed consent with full understanding of this clinical trial
8. A healthy person who does not have clinically significant findings in the clinical laboratory test, vital signs, and physical examination

Exclusion Criteria:

1. Allergic to beans, lidocaine or medical devices which used in this clinical trial (sterile oil pan, alcohol swab, grid pad, needle, etc.)
2. Central, endocrine, or hereditary obesity (BMI 35kg/m^2 or more)
3. History of any treatment (orthognathic surgery, suction lipectomy, PPC injection) in the neck or chin area
4. Inflammation, scars or surgery on the injection area
5. history of dysphagia or current symptoms of dysphagia
6. Clinical laboratory tests and electrocardiogram results performed during screening visit are clinically significant abnormal factors.

   * Total Cholesterol > 250 mg/dl, LDL-C > 160 mg/dL, TG > 200 mg/dL
   * AST, ALT, γ-GT > 2x the upper limit of the normal range
   * CK > 2.5 times the upper limit of the normal range
   * eGFR (MDRD) <60 ml/min/1.73m2,MDRD=175*Scr[exp(-1.154)]*AGE[exp(-0.203)]*[0.742 (for women)]
7. Positive results of virus tests (HBV, HCV, HIV) performed during screening visit
8. Positive results of syphilis test (RPR) performed during screening visit
9. unable to participate by the tester due to serious medical or psychiatric diseases falling under the following conditions

   ① Respiratory diseases: People who need to take daily medication such as asthma, chronic obstructive pulmonary disease (COPD), active tuberculosis, latent tuberculosis under treatment, etc
   * Severe cardiovascular disease: congestive heart failure, coronary artery disease, myocardial infarction, uncontrolled high blood pressure, myocarditis, pericarditis, etc

     * Neurological disorders: Epilepsy, Seizure (within 3 years prior to clinical trial medication), stroke, encephalopathy, Guillain-Barre syndrome, encephalomyelitis, transverse spondylitis, etc

       * Malignant tumor history within 5 years before IP administration of clinical trial drugs (except for basal cell and squamous cell carcinoma) ⑤ Autoimmune hypothyroidism and autoimmune diseases including psoriasis ⑥ Immunodeficiency disease ⑦Other diseases such as the hepatobiliary, kidney, endocrine system, urology, and musculoskeletal system that were determined to be clinically significant by PI
10. Diagnosis of heart disease (cardiac failure, unstable angina, myocardial infarction) or stroke within 6 months before screening
11. Administration of anticoagulants or anticoagulants with a history of platelet-related or hemorrhagic diseases or a history of severe bleeding or bruising after previous subcutaneous injection
12. history of systemic hives within 5 years before IP administration
13. history of genetic or idiopathic vascular neuropathy
14. organ or bone marrow transplantation
15. suspected of drug abuse or alcohol abuse or has a history within six months before IP administration
16. uses immunosuppressants and immunomodulators or chronically uses steroids within 6 months before IP administration

    ① Immunosuppressants and regulators : : Azathioprine, Cyclosporine, Interferon, G-CSF, Tacrolimus, Everolimus, Sirolimus, Cyclophosphamide, 6-Mercaptopurine, Methotrexate, Rapamycin, Leflunomide etc.

    ② Systemic steroids: If a dose of more than 10 mg/day based on Prednisolone is used for more than 14 consecutive days (but steroids, nasal sprays, inhalants and eye drops are allowed regardless of the volume of use)
17. history of dependent administration of psychotropic drugs or narcotic painkillers within 6 months before IP administration or who is mentally ill or in a social condition that is difficult to comply with clinical trial procedures at the discretion of PI
18. taken any ETC drug or herbal medicine within two weeks prior to the first dose date, or who has taken any general drug (OTC drug) or fish oil preparation (Omega3) within one week (but may participate in clinical trials if other conditions are reasonable)
19. continue to drink (over 21 units/week, 1 unit = 10 g of pure alcohol) or who cannot abstain from drinking during the clinical trial
20. Smokers (in some cases, smoking up to 10 cigarettes/day is acceptable at the discretion of PI)
21. have participated in other clinical trials (including live trials) within 6 months before IP administration
22. has been administered immunoglobulin or blood-derived drugs within three months before IP administration, or a person who has plans to administer them during the clinical trial period
23. has donated the following blood prior to the first date of administration

    - Whole blood; 2 months; component blood donation; within 1 month
24. a pregnant or lactating woman
25. has determined that PI is not eligible for this clinical trial due to other reasons

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Safety- Number of adverse event, incidence of adverse event | IP treatment~ the end visit of the clinical trial : 28 day
  AE to the localized injection area or total body)

SECONDARY OUTCOMES:
Pharmacokinetics- Cmax of DLPC(IPsurface substances) | baseline IP treatment, Amount of change
  Peak Plasma Concentration(Cmax), Tmax etc. of DLPC(IP surface substances)
Pharmacokinetics- AUC of DLPC(IPsurface substances) | baseline IP treatment, Amount of change
  Area under the plasma concentration versus time curve(AUC) of DLPC(IPsurface substances)

CONTACTS AND LOCATIONS:
Overall Officials: Jae Yong Chung, M.D.,Ph.D, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee HJ, Jiang X, Abd El-Aty AM, Jeong JH, Chung JY. Phase 1 study of AYP-101 (soybean phosphatidylcholine): safety, pharmacokinetics, and lipid profile effects for reducing submental fat. Lipids Health Dis. 2024 Dec 28;23(1):426. doi: 10.1186/s12944-024-02387-4. PMID 39732703